CLINICAL TRIAL: NCT06486506
Title: Proximal Femur Reconstruction Following Resection of Primary Bone Tumors: Analysis of the Clinical and Radiographic Results
Acronym: ProFemuRe
Status: Recruiting | Type: Observational
Sponsor: Costantino Errani (Other)
Responsible Party: Sponsor-Investigator, Costantino Errani, Principal Investigator, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: ProFemuRe
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Bone Tumor; Bone Cancer
Keywords: Proximal Femur Reconstruction; primary bone tumors; imaging
MeSH Terms: conditions — Bone Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients: Male and female patients surgically treated with an oncological reconstruction of the proximal femur at Rizzoli Orthopaedic Institute between 01/01/1991 and 31/12/2023
  Interventions: Other: Analysis

INTERVENTIONS:
Other: Analysis — Analysis and review of imaging and clinical data

SUMMARY:
From the archives of the Rizzoli institute all the patients (approximately 150 patients) undergoing oncological reconstruction of proximal femur from 01/01/1991 to 31/12/2023.

A review will be made from the medical records, radiological imaging, and histological data of these patients

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients surgically treated with an oncological reconstruction of the proximal femur at Rizzoli Orthopaedic Institute between 01/01/1991 and 31/12/2023
* Age: 18-90 years old (at the time of primary surgery)
* Diagnosis of bone sarcoma
* Patients with available clinical and imaging data

Exclusion Criteria:

* At least one inclusion criterion not met

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male and female patients surgically treated with an oncological reconstruction of the proximal femur at Rizzoli Orthopaedic Institute between 01/01/1991 and 31/12/2023
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
longevity of the reconstruction | At baseline (Day 0)
  evaluation of the longevity of the reconstruction, meaning reconstruction failure-free survival after surgery

SECONDARY OUTCOMES:
Musculoskeletal tumour society (MSTS) functional evaluation | at baseline (day 0)
  The MSTS questionnaire consists of six domains, each scored on a scale from 0 to 5, with a higher score indicating better function.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Itituto Ortopedico Rizzoli, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tobey D, Wing C, Calkins T, Heck RK. The Use of Proximal Femur Replacement for the Management of Oncologic Lesions in the Proximal Femur: A Review. Orthop Clin North Am. 2023 Jan;54(1):23-35. doi: 10.1016/j.ocl.2022.08.006. Epub 2022 Oct 23. PMID 36402508
- [Background] Menendez LR, Ahlmann ER, Kermani C, Gotha H. Endoprosthetic reconstruction for neoplasms of the proximal femur. Clin Orthop Relat Res. 2006 Sep;450:46-51. doi: 10.1097/01.blo.0000229332.91158.05. PMID 16906093